CLINICAL TRIAL: NCT05782556
Title: Transjugular Intrahepatic Portosystemic Shunt (TIPS) for the Treatment of Portal Hypertension: an Observational Study
Brief Title: Freiburg TIPS Registry
Acronym: FRETIR
Status: Recruiting | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, PD Dr. Dominik Bettinger, MD, University Hospital Freiburg
Other Study IDs: FRETIR01
Record Dates: First submitted 2023-03-10; First posted 2023-03-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Non-Cirrhotic Portal Hypertension; Budd Chiari Syndrome; Portal Vein Thrombosis; Portal Systemic Shunt
Keywords: Liver cirhosis; Transjugular intrahepatic portosystemic shunt; Non-Cirrhotic Portal Hypertension; Prognosis; Outcome
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Budd-Chiari Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Serum, plasma, peripheral blood mononuclear cell (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients allocated to implantation of a transjugular intrahepatic portosystemic shunt (TIPS): Patients allocated to implantation of a transjugular intrahepatic portosystemic shunt (TIPS) due to cirrhotic and non-cirrhotic portal hypertension
  Interventions: Device: Implantation of a transjugular intrahepatic portosystemic shunt (TIPS)

INTERVENTIONS:
Device: Implantation of a transjugular intrahepatic portosystemic shunt (TIPS) — For TIPS implantation, a transjugular approach is used in all patients and a puncture needle was advanced into a hepatic vein. Puncture of the portal vein is performed using ultrasound guidance followed by portography after successful puncture of the portal vein. Further, the parenchymal tract isdilated and the stent graft is placed. Before and after TIPS implantation, portal venous and central venous pressures are measured to calculate the porto-systemic pressure gradient

SUMMARY:
Patients with clinically significant portal hypertension allocated to implantation of a transjugular intrahepatic portosystemic shunt (TIPS) at the Department of Medicine II of the University Medical Center Freiburg, Germany will be offered to participate in this prospective observational trial.

Clinical and laboratory as well as outcome parameters will be assessed before and within the first 12 months after TIPS implantation following a regular follow-up schedule with clinical visits at the University Medical Center Freiburg. During follow-up visits, serum/plasma samples and peripheral blood mononuclear cells (PBMC) are collected and stored in a associated biobank.

DETAILED DESCRIPTION:
Patients with clinically significant cirrhotic and non-cirrhotic portal hypertension who are allocated to implantation of a transjugular intrahepatic portosystemic shunt (TIPS) can be included in this observational study. Further patients who have been treated between 01/01/2005 and the start of the prospective part of this study (01/01/2023) will be included retrospectively in this registry.

Patients who are allocated to TIPS implantation will be recruited the day before TIPS implantation. Detailled patient characteristics, epidemiologic, clinical, imaging and laboratory parameters will be assessed and included in an electronic database. Further, interventional data of TIPS implantation will be included in the database.

Apart from these data, patients will be asked to participate in biobank sampling including serum/plasma and peripheral blood mononuclear cells (PBMC) samples from the peripheral veins and from the liver and portal vein that will be taken during TIPS implantation.

All patients recruited in this registry will be followed-up for at least 12 months with regular visits 3, 6 and 12 months after TIPS implantation.

Outcome parameters including development of post-TIPS hepatic encephalopathy, acute- on chronic liver failure (ACLF), infections, recurrence of clinically significant portal hypertension, need for TIPS revision and death and liver transplantation will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients allocated to TIPS implantation due to clinically significant cirrhotic and non-cirrhotic portal hypertension

Exclusion Criteria:

* Withdrawal of written informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients allocated to TIPS implantation due to clinically significant cirrhotic and non-cirrhotic portal hypertension will be included in this study.In summary, patients with the folowing conditions can be included:
  * liver cirrhosis and indication for TIPS implantation (pre-emptive TIPS or rescue TIPS in case of varical bleeding, secondary prophylaxis of varical bleeding, recurrent or refractory ascites, TIPS before surgery)
  * non-cirrhotic portal vein thrombosis
  * Budd-Chiari syndrome
  * porto-sinusoidal vascular disease
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2034-06-30 (Estimated)

PRIMARY OUTCOMES:
Transplantation-free survival | 01/01/2023-31/12/2033
  Time from study inclusion to death or liver transplantation

SECONDARY OUTCOMES:
Time to development of post-TIPS hepatic encephalopathy | 01/01/2023-31/12/2033
  Time from study inclusion to development of post-TIPS hepatic encephalopathy
Time to development of post-TIPS acute- on chronic liver failure (ACLF) | 01/01/2023-31/12/2033
  Time from study inclusion to development of post-TIPS ACLF
Time to need for TIPS revision | 01/01/2023-31/12/2033
  Time from study inclusion to need for TIPS revision
Prevalence of osteoporosis in patients with TIPS implantation | 01/01/2023-31/12/2033
  Osteoporosis is assessed by DXA measurement
Impact of osteoporosis on prognosis and decompensating events after TIPS | 01/01/2023-31/12/2033
  Osteoporosis is assessed by DXA measurement. Bone density will be correlated with prognosis and decompensating events.
Prevalence of sarcopenia in patients with TIPS implantation | 01/01/2023-31/12/2033
  Sarcopenia is assessed by computed tomography.
Impact of sarcopenia on prognosis and decompensating events after TIPS | 01/01/2023-31/12/2033
  Sarcopenia is assessed by computed tomography and is correlated with prognosis and the development of decompensating events after TIPS
Time to development of post-TIPS infections/sepsis | 01/01/2023-31/12/2033
  Time from study inclusion to development of post-TIPS infections/sepsis
Periinterventional complications | 01/01/2023-31/12/2033
  Periinterventional complications (infections, bleeding, biliary injury) are assessed during the intervention. These complications are documented in the report of the intervention and are assessed systematically.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Bettinger, MD, Principal Investigator — University Hospital Freiburg
Locations (1):
- University Medical Center Freiburg, Department of Medicine II, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heger LA, Chang J, Rohrer C, Reincke M, Eyth A, Sturm L, Schultheiss M, Maier A, Meyer C, Jansen C, Graf K, Ozturk C, Schneider F, Trebicka J, Westermann D, Thimme R, Grundmann S, Praktiknjo M, Bettinger D. Right Ventricular Contractility Predicts Clearance of Ascites After Transjugular Intrahepatic Portosystemic Shunt. Liver Int. 2025 Dec;45(12):e70422. doi: 10.1111/liv.70422. PMID 41204773
- See also: Homepage Interventional Hepatology University Medical Center Freiburg — http://www.uniklinik-freiburg.de/medizin2/forschung/klinische-forschung/ag-schultheissbettinger.html